CLINICAL TRIAL: NCT00225784
Title: A Phase II Trial of Cetuximab, Radiotherapy and Twice Weekly Gemcitabine in Patients With Adenocarcinoma of the Pancreas
Brief Title: Cetuximab, Radiotherapy and Twice Weekly Gemcitabine to Treat Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DMS 0432
Record Dates: First submitted 2005-09-22; First posted 2005-09-26 (Estimated); Results first posted 2013-04-18 (Estimated); Last update posted 2014-07-16 (Estimated); Status verified 2011-10

CONDITIONS: Pancreatic Cancer
Keywords: Stage I, II, III pancreatic adenocarcinoma; Radiographically measurable disease
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Cetuximab; Gemcitabine; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cetuximab, Gemcitabine, RT (Experimental): weekly cetuximab, twice-weekly gemcitabine and intensity modulated radiotherapy
  Interventions: Drug: Cetuximab/Gemcitabine; Procedure: Radiotherapy

INTERVENTIONS:
Drug: Cetuximab/Gemcitabine — Once weekly Cetuximab, twice weekly Gemcitabine for six weeks
  Other Names: Erbitux
Procedure: Radiotherapy — Daily radiotherapy for 28 days

SUMMARY:
This study is designed to establish the safety and efficacy of a combination of Erbitux (cetuximab)/Gemzar (gemcitabine)/radiation in patients with pancreatic cancer.

DETAILED DESCRIPTION:
The study treatment for this protocol is

* Loading dose of Cetuximab 400 mg/m2
* Weekly Cetuximab 250 mg/m2
* Bi-weekly Gemcitabine 50 mg/m2
* Daily Radiation for 28 fractions
* CT scan four weeks after completion of treatment
* Evaluation by surgeon for resectability

ELIGIBILITY:
Inclusion Criteria:

* Histologic proof of pancreatic adenocarcinoma
* Clinical stage I, II, or III disease
* Radiographically measurable disease
* Tumor tissue for epidermal growth factor receptor (EGFR) status by immunohistochemistry
* Signed protocol consent
* Karnofsky performance status of at least 70%
* Age > or = to 18 years
* Patients must either not be of child bearing potential or have a negative pregnancy test within 72 hours of treatment.
* Absolute neutrophil count (ANC) > 1500; platelets > 100,000/ul.
* Creatinine < 1.5 x upper limit of normal (ULN)
* Bilirubin < 1.5 x ULN; AST < 2.5 x ULN.

Exclusion Criteria:

* Acute hepatitis or known HIV
* Active or uncontrolled infection
* Significant history of cardiac disease
* Prior therapy which affects or targets the EGF pathway
* Prior severe infusion reaction to a monoclonal antibody
* Any concurrent chemotherapy not indicated in the study protocol or any other investigational agents
* Any previous chemotherapy or abdominal or pelvic radiotherapy
* No prior malignancy is allowed except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or malignancy for which the patient has been disease free for five years.
* Any severe pre-existing medical or psychiatric condition, which, in the opinion of the attending physician, will interfere with safe and appropriate treatment and follow-up on study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2005-02; Primary Completion 2010-02 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: J Marc Pipas, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a single-institution study of weekly cetuximab, twice-weekly gemcitabine and intensity modulated radiotherapy in patients with pancreatic ductal adenocarcinoma conducted at Dartmouth-Hitchcock.
Groups:
- Cetuximab, Gemcitabine, Radiotherapy: Weekly cetuximab, twice-weekly gemcitabine and intensity modulated radiotherapy
Period: Overall Study
Arm/Group | Cetuximab, Gemcitabine, Radiotherapy
Started | 37
Completed | 33
Not Completed | 4

BASELINE CHARACTERISTICS:
Groups:
- Cetuximab/Gemcitabine/Radiotherapy: weekly cetuximab, twice-weekly gemcitabine and intensity modulated radiotherapy
Arm/Group | Cetuximab/Gemcitabine/Radiotherapy
Number analyzed (Participants) | 37
Age, Continuous [Mean (Inter-Quartile Range); unit: years]
  Between 18 and 65 years | 54.7 [39 to 65]
  >=65 years | 73.1 [67 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 16

OUTCOME MEASURES:

1. Primary Outcome: Objective Response of Tumor by RECIST 1.0 Criteria
Description: Per RECIST Criteria (v. 1.0) and assessed by CT scan: Complete Response (CR), disappearance of all target lesions; Partial Response (PR), >=30% decrease in sum of the longest diameter (SLD)of target lesions at baseline; Progressive Disease (PD), >=20% increase in the SLD of target lesions at baseline; Stable Disease (SD), Neither sufficient decrease in SLD to qualify for PR nor sufficient increase in SLD to qualify for PD.
Time Frame: one month post-therapy
Population: Completion of treatment
Measure: Number; unit: participants
Arm/Group | Cetuximab, Gemcitabine, Radiotherapy
Number analyzed (Participants) | 33
participants
  partial response | 10
  stable disease | 20
  progressive disease | 3

2. Secondary Outcome: Number of Participants Assessed for Adverse Events
Description: Adverse events assessed using Common Terminology Criteria for Adverse Events version 3.0
Time Frame: Participants were followed during treatment and for 30 days after completion of treatment
Population: All participants were evaluated for toxicity.
Measure: Number; unit: participants
Groups:
- Cetuximab, Gemcitabine, Radiotherapy: Weekly cetuximab twice-weekly gemcitabine plus intensity modulated radiotherapy.
Arm/Group | Cetuximab, Gemcitabine, Radiotherapy
Number analyzed (Participants) | 37
participants | 37

3. Secondary Outcome: Number of Participants Determined to be Resectable (Eligible for Surgery)After Completion of Therapy
Description: Tumor resectability is based on CT scan and as defined by the American Hepato-Pancreato-Biliary Association Convened Consensus Conference on Resectable and Borderline Resectable Pancreatic Cancer (Callery MP, et al. Ann Surg Oncol 2009; 16:1727-1733): no evidence of superior mesenteric vein (SMV) or portal vein (PV)abutment, distortion, tumor thrombus, or venous encasement, and clear fat planes around celiac axis (CA), hepatic artery (HA), and superior mesenteric artery (SMA).
Time Frame: 1 month after completion of treatment
Population: Surviving participants who completed therapy and were determined to be resectable.
Measure: Number; unit: participants
Arm/Group | Cetuximab, Gemcitabine, Radiotherapy
Number analyzed (Participants) | 33
participants | 26

4. Secondary Outcome: Role of Epidermal Growth Factor Receptor (EGFR) Status in Response to Treatment.
Description: Tumor was assessed for EGFR status by immunohistochemistry. EGFR positive and EGRF negative tumor types were evaluated and compared for response to treatment.
Time Frame: One month post-therapy
Population: All EGFR (-) subjects who completed therapy were evaluated.
Measure: Number; unit: percent
Groups:
- Cetuximab, Gemcitabine, Radiotherapy in EGFR (-) Tumors: Percentage of response to weekly cetuximab, twice-weekly gemcitabine and intensity modulated radiotherapy in patients with EGFR negative tumors.
- Cetuximab, Gemcitabine, Radiotherapy in EGFR (+) Tumors: Percentage of response to weekly cetuximab, twice-weekly gemcitabine and intensity modulated radiotherapy in patients with EGFR positive tumors.
Arm/Group | Cetuximab, Gemcitabine, Radiotherapy in EGFR (-) Tumors | Cetuximab, Gemcitabine, Radiotherapy in EGFR (+) Tumors
Number analyzed (Participants) | 9 | 24
percent | 33 | 29

5. Secondary Outcome: Disease-Free Survival After Therapy
Description: Time to disease progression after therapy.
Time Frame: Five years post treatment
Population: All evaluable participants who completed treatment, and had confirmed progression of disease.
Measure: Median (Full Range); unit: months
Arm/Group | Cetuximab, Gemcitabine, Radiotherapy
Number analyzed (Participants) | 28
months | 9.1 [2 to NA] — Partipants did not all reach endpoint.

6. Secondary Outcome: Overall Length of Survival After Therapy
Description: Length of survival after therapy in all participants enrolled.
Time Frame: Five years post treatment
Population: All participants enrolled regardless of evaluability for primary outcome measure.
Measure: Median (Full Range); unit: months
Arm/Group | Cetuximab, Gemcitabine, Radiotherapy
Number analyzed (Participants) | 37
months | 17.3 [2 to NA] — Not all participants evaluated reached end point.

7. Secondary Outcome: Pattern of Failure After Therapy
Description: Local recurrence, distant recurrence, or both.
Time Frame: Five years post treatment
Population: All participants who completed treatment and underwent resection
Measure: Number; unit: participants
Arm/Group | Cetuximab, Gemcitabine, Radiotherapy
Number analyzed (Participants) | 25
participants
  number of participants with local recurrence only | 2
  number of ppts. with local and distant recurrence | 1
  number of ppts. with distant disease recurrence | 17
  number of ppts. without recurrence or unknown | 5

ADVERSE EVENTS:
Arm/Group | Cetuximab/Gemcitabine/Radiotherapy
Serious Adverse Events (participants affected / at risk) | 22/33
Other Adverse Events (participants affected / at risk) | 3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cetuximab/Gemcitabine/Radiotherapy (N=33)
CNS Ischemia (Nervous system disorders) | 2 (2)
Anemia (Investigations) | 1 (1)
Gastrointestinal disorder - stent obstruction (Gastrointestinal disorders) | 8 (8) — Stent obstruction is common in patients with pancreatic cancer.
Deep vein thrombosis (Vascular disorders) | 2 (2)
Fatigue (General disorders) | 4 (4)
Gastritis/GI Bleed (Gastrointestinal disorders) | 5 (5)
Hematoma subdural (Nervous system disorders) | 1 (1) — This was related to a traumatic event, not to treatment.
Nausea/Vomiting (Gastrointestinal disorders) | 9 (16)
Pain - gouty arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 22 (34) — Of the 22 patients experiencing Grade 3 neutropenia, only one developed neutropenic fever requiring hospitalization. The other 21 were managed in an outpatient setting.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk (number of events):
Term (organ system) | Cetuximab/Gemcitabine/Radiotherapy
Anaphylaxtic reaction to erbitux (Immune system disorders) | 3/37 (3)

LIMITATIONS AND CAVEATS:
Our study suffers limitations common to single institution trials, namely small patient numbers and selection bias. Our cohort of subjects is too small to adequately assess the effect of tumor EGFR and KRAS status on outcome.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No